CLINICAL TRIAL: NCT05429970
Title: Perioperative Stress Reduction in Ovarian Cancer (PRESERVE Trial)-A Prospective Randomized Pilot Study
Brief Title: A Study Comparing Perioperative Stress Reduction vs. Standard of Care in Ovarian Cancer (PRESERVE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-049
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer; Ovarian Carcinoma; Stage II Ovary Cancer; Stage II Ovarian Cancer; Stage III Ovary Cancer; Stage III Ovarian Cancer; Stage IV Ovary Cancer; Stage IV Ovarian Cancer; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Stage II Fallopian Tube Cancer; Stage III Fallopian Tube Cancer; Stage IV Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: ovarian cancer; propranolol; etodolac; MBRT; mind-body resilience training; music therapy; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Music Therapy; Propranolol; Etodolac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PSRB (Experimental): Participants will receive mind-body resilience training/MBRT, music therapy, propranolol and etodolac pre and post operatively. Postoperative Psychological Interventions may occur between POD 1-7 if needed.
  Interventions: Behavioral: Mind-body resilience training; Behavioral: Music therapy; Drug: Propranolol; Drug: Etodolac
- Standard of Care (No Intervention): Participants will receive usual care (study interventions not specifically recommended)

INTERVENTIONS:
Behavioral: Mind-body resilience training — MBRT is a meditation technique used to achieve relaxation)
  Other Names: MBRT
  Arms: PSRB
Behavioral: Music therapy — Music listening was found, in multiple trials, to significantly reduce self-reported anxiety, physiologic indicators of anxiety, and/or sedation requirements
  Arms: PSRB
Drug: Propranolol — Propranolol 20 mg PO BID (for 21 consecutive days), Propranolol 10mg PO BID (for 3 consecutive days POD 14-16)
  Arms: PSRB
Drug: Etodolac — Etodolac 400 mg PO BID (for 21 consecutive days)
  Arms: PSRB

SUMMARY:
The purpose of this study is to see if propranolol and etodolac along with mind-body resilience training/MBRT and music therapy help participants who are experiencing physiological stress before, during, and after primary debulking surgery/PDS or IDS and also if it's better than the standard-of-care approach (no intervention for reducing stress).

ELIGIBILITY:
Inclusion Criteria:

* Advanced (stage II-IV) epithelial ovarian, fallopian tube, or primary peritoneal carcinoma diagnosed on the basis of imaging, CA125, and clinical assessment
* Scheduled to undergo exploratory laparotomy and PDS or IDS
* Scheduled for surgery with at least 10 days of lead time, to allow the participant to take the β-blocker and COX2 inhibitor 7 days preoperatively
* Age ≥18 years
* ASA score of 1 to 3
* Ability to understand the study objectives and procedures, comply with the protocol, and provide informed consent

Exclusion Criteria:

* Chronic treatment with any β-blocker or COX inhibitor
* Contraindication for β-blocker therapy (asthma, second- or third-degree atrioventricular block, sinus bradycardia, sick sinus syndrome, right-sided heart failure, pheochromocytoma, peripheral vascular disease)
* Contraindication for COX2 inhibitor therapy (renal failure [creatinine level >1.5 mg/dL], significant liver failure [known cirrhosis, bilirubin level >2], active peptic disease), or current use of oral anticoagulant)
* Contraindication for regional epidural anesthesia
* Chronic autoimmune disease
* Active infection
* Pregnant
* Minimally invasive procedure
* Participation in another clinical trial that interferes with this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants successfully completing over 80% of the bundled interventions | 21 days after surgical procedure
  The primary objective of this study is to investigate the feasibility of implementing a multimodal PSRB in women undergoing PDS or IDS for advanced EOC. This will be measured as number of patients successfully completing over 80% of the bundled interventions, including a preoperative integrative medicine session, postoperative integrative medicine session, total intravenous anesthesia on day of surgery, and perioperative beta blocker and COX2 inhibitor

CONTACTS AND LOCATIONS:
Overall Officials: Kara Long Roche, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org